CLINICAL TRIAL: NCT05793229
Title: Exploration of Frailty Trajectories and Their Association With Health Outcomes in Elderly Gastric Cancer Survivors Undergoing Radical Gastrectomy: a Prospective Longitudinal Observation Study
Brief Title: Frailty Trajectories and Their Association With Health Outcomes
Status: Completed | Type: Observational
Sponsor: Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Xueyi Miao, Principal Investigator, Nanjing Medical University
Other Study IDs: Nanjing Medical University
Record Dates: First submitted 2023-03-19; First posted 2023-03-31 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Frailty Syndrome
MeSH Terms: conditions — Frailty | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- improving frailty: Class 1
  Interventions: Other: observation
- maintaining frailty: Class 2
  Interventions: Other: observation
- deteriorating frailty: Class 3
  Interventions: Other: observation

INTERVENTIONS:
Other: observation — observation

SUMMARY:
Frailty is common in gastric cancer survivors and seriously affects their prognosis. Multiple longitudinal follow-up assessment of frailty could provide a better understanding of the frailty change of individuals. Our aims were to identify the longitudinal trajectories of frailty and estimate their association with health outcomes in elderly gastric cancer survivors.

DETAILED DESCRIPTION:
Our study suggested the significant heterogeneity in frailty trajectories among elderly gastric cancer survivors, and that different trajectories had different effects on health outcomes. Our results infer the necessity for prevention strategies in elderly gastric cancer survivors to manage heterogeneous frailty trajectories.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with gastric cancer by endoscopy or pathology;
* received radical gastrectomy the first time;
* aged ≥60 years;
* been able to communicate simply in writing and verbal;
* completed the data collection of all follow-up points.

Exclusion Criteria:

* received radiotherapy or chemotherapy before surgery;
* had other sites of malignant tumors;
* complicated with severe heart, liver, lung and renal insufficiency;
* had physical disability.

Min Age: 60 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Elderly patients with gastric cancer who attended a tertiary care hospital in China from March 2021 to October 2021 were selected for the study.
Sampling Method: Non-Probability Sample
Enrollment: 381 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
quality of life (QOL) | at 1-year after surgery
  used EORTC QLQ-STO22 to assess.
disability | at 1-year after surgery
  used Elderly Disability Assessment Scale to assess.
1-year hospital readmissions | at 1-year after surgery
  captured from medical records.
total costs | at 1-year after surgery
  captured from medical records.

CONTACTS AND LOCATIONS:
Locations (1):
- Xueyi Miao, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided